CLINICAL TRIAL: NCT03474107
Title: An Open-Label, Randomized Phase 3 Study to Evaluate Enfortumab Vedotin vs Chemotherapy in Subjects With Previously Treated Locally Advanced or Metastatic Urothelial Cancer (EV-301)
Brief Title: A Study to Evaluate Enfortumab Vedotin Versus (vs) Chemotherapy in Subjects With Previously Treated Locally Advanced or Metastatic Urothelial Cancer (EV-301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7465-CL-0301; 2017-003344-21 (EudraCT Number); jRCT2080224027 (Registry Identifier: jRCT); 2024-517571-20-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT04136808 (Approved for marketing)
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Ureteral Cancer; Urothelial Cancer; Bladder Cancer
Keywords: antibody drug conjugate; enfortumab vedotin (EV); ASG-22ME; ASG-22CE; urothelial cancer
MeSH Terms: conditions — Ureteral Neoplasms; Urinary Bladder Neoplasms | interventions — enfortumab vedotin; Docetaxel; vinflunine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Enfortumab Vedotin 1.25 mg/kg (Experimental): Participants received 1.25 milligrams per kilogram (mg/kg) of body weight enfortumab vedotin by intravenous infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
  Interventions: Drug: Enfortumab Vedotin
- Arm B: Chemotherapy (Active Comparator): Participants received either 75 milligrams per square meter (mg/m^2) docetaxel by IV infusion over approximately 1 hour or 320 mg/m^2 vinflunine by IV infusion over approximately 20 minutes or 175 mg/m^2 paclitaxel by IV infusion over approximately 1 hour on day 1 of every 21-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
  Interventions: Drug: Docetaxel; Drug: Vinflunine; Drug: Paclitaxel
- Cross-over Extension (COE) (Experimental): Eligible participants from chemotherapy arm who met the criteria for COE will receive 1.25 mg/kg of body weight enfortumab vedotin by intravenous infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle until discontinuation criteria is met.
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Enfortumab Vedotin — Intravenous infusion
  Other Names: ASG-22ME; ASG-22CE
  Arms: Arm A: Enfortumab Vedotin 1.25 mg/kg; Cross-over Extension (COE)
Drug: Docetaxel — Intravenous infusion
  Arms: Arm B: Chemotherapy
Drug: Vinflunine — Intravenous infusion
  Arms: Arm B: Chemotherapy
Drug: Paclitaxel — Intravenous infusion
  Arms: Arm B: Chemotherapy

SUMMARY:
The purpose of this study was to compare the overall survival (OS) of participants with locally advanced or metastatic urothelial cancer treated with enfortumab vedotin (EV) to the OS of participants treated with chemotherapy.

This study compared progression-free survival on study therapy (PFS1); the overall response rate (ORR) and the disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 of participants treated with EV to participants treated with chemotherapy.

In addition, this study evaluated the duration of response (DOR) per RECIST V1.1 of EV and chemotherapy and assessed the safety and tolerability of EV, as well as, the quality of life (QOL) and Patient Reported Outcomes (PRO) parameters.

DETAILED DESCRIPTION:
Japan PMDA has approved enfortumab vedotin (Padcev) for the treatment of advanced urothelial cancer. The study will continue as a post marketing study in Japan.

Participants considered an adult according to local regulation at the time of obtaining informed consent participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is legally an adult according to local regulation at the time of signing informed consent.
* Subject has histologically or cytologically confirmed urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Subjects with urothelial carcinoma (transitional cell) with squamous differentiation or mixed cell types are eligible.
* Subject must have experienced radiographic progression or relapse during or after a checkpoint inhibitor (CPI) (anti-programmed cell death protein 1 (PD1) or anti-programmed death-ligand 1 (PD-L1)) for locally advanced or metastatic disease. Subjects who discontinued CPI treatment due to toxicity are eligible provided that the subjects have evidence of disease progression following discontinuation. The CPI need not be the most recent therapy. Subjects for whom the most recent therapy has been a non-CPI based regimen are eligible if the subjects have progressed/relapsed during or after the subjects most recent therapy. Locally advanced disease must not be amenable to resection with curative intent per the treating physician.
* Subject must have received a platinum containing regimen (cisplatin or carboplatin) in the metastatic/locally advanced, neoadjuvant or adjuvant setting. If platinum was administered in the adjuvant/neoadjuvant setting subject must have progressed within 12 months of completion.
* Subject has radiologically documented metastatic or locally advanced disease at baseline.
* An archival tumor tissue sample should be available for submission to central laboratory prior to study treatment. If an archival tumor tissue sample is not available, a fresh tissue sample should be provided. If a fresh tissue sample cannot be provided due to safety concerns, enrollment into the study must be discussed with the medical monitor.
* Subject has ECOG PS of 0 or 1
* The subject has the following baseline laboratory data:

  * absolute neutrophil count (ANC) ≥ 1500/mm3
  * platelet count ≥ 100 × 10^9/L
  * hemoglobin ≥ 9 g/dL
  * serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease
  * creatinine clearance (CrCl) ≥ 30 mL/min as estimated per institutional standards or as measured by 24 hour urine collection (glomerular filtration rate [GFR] can also be used instead of CrCl)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 3 x ULN for subjects with liver metastases
* Female subject must either:

  * Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for at least 6 months after the final study drug administration, and have a negative urine or serum pregnancy test within 7 days prior to Day 1 (Females with false positive results and documented verification of negative pregnancy status are eligible for participation), and if heterosexually active, agree to consistently use a condom plus 1 form of highly effective birth control per locally accepted standards starting at screening and throughout the study period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed or donate ova starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
* A sexually active male subject with female partner(s) who is of childbearing potential is eligible if:

  * Agrees to use a male condom starting at screening and continue throughout the study treatment and for at least 6 months after final study drug administration. If the male subject has not had a vasectomy or is not sterile as defined below the subjects female partner(s) is utilizing 1 form of highly effective birth control per locally accepted standards starting at screening and continue throughout study treatment and for at least 6 months after the male subject receives final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to abstinence or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for at least 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment in present study.

Inclusion Criteria for COE:

* Subject is eligible for the COE if they continue to meet all inclusion criteria from the main protocol in addition to the following when the patient is evaluated for eligibility to participate in the COE portion of the study:
* Institutional review board (IRB)/ independent ethics committee (IEC) approved written COE informed consent and privacy language as per national regulations (e.g., health insurance portability and accountability act [HIPAA] Authorization for US sites) must be obtained from the subject prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
* Subject was randomized to Arm B and is either currently on study treatment or has discontinued study treatment due to intolerance, AE or progression of disease and has not started a new systemic anticancer treatment.

Exclusion Criteria:

* Subject has preexisting sensory or motor neuropathy Grade ≥ 2.
* Subject has active central nervous system (CNS) metastases. Subjects with treated CNS metastases are permitted on study if all the following are true:

  * CNS metastases have been clinically stable for at least 6 weeks prior to screening
  * If requiring steroid treatment for CNS metastases, the subject is on a stable dose ≤ 20 mg/day of prednisone or equivalent for at least 2 weeks
  * Baseline scans show no evidence of new or enlarged brain metastasis
  * Subject does not have leptomeningeal disease
* Subject has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery). Subject with ≤ Grade 2 immunotherapy-related hypothyroidism or panhypopituitarism may be enrolled when well-maintained/controlled on a stable dose of hormone replacement therapy (if indicated). Subjects with ongoing ≥ Grade 3 immunotherapy-related hypothyroidism or panhypopituitarism are excluded. Subjects with ongoing immunotherapy related colitis, uveitis, or pneumonitis or subjects with other immunotherapy related AEs requiring high doses of steroids (> 20 mg/day of prednisone or equivalent) are excluded.
* Subject has prior treatment with EV or other monomethyl auristatin E (MMAE)-based Antibody drug conjugates (ADCs).
* Subject has received prior chemotherapy for urothelial cancer with all available study therapies in the control arm (i.e., both prior paclitaxel and docetaxel in regions where vinflunine is not an approved therapy, or prior paclitaxel, docetaxel and vinflunine in regions where vinflunine is an approved therapy).
* Subject has received more than 1 prior chemotherapy regimen for locally advanced or metastatic urothelial cancer, including chemotherapy for adjuvant or neo-adjuvant disease if recurrence occurred within 12 months of completing therapy. The substitution of carboplatin for cisplatin does not constitute a new regimen provided no new chemotherapeutic agents were added to the regimen.
* Subject has history of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Subjects with nonmelanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Subject is currently receiving systemic antimicrobial treatment for viral, bacterial, or fungal infection at the time of first dose of EV. Routine antimicrobial prophylaxis is permitted.
* Subject has known active Hepatitis B (e.g., hepatitis B surface antigen (HBsAg) reactive) or active hepatitis C (e.g., hepatitis C virus (HCV) Ribonucleic Acid (RNA) [qualitative] is detected).
* Subject has known history of human immunodeficiency virus (HIV) infection (HIV 1 or 2).
* Subject has documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study drug.
* Subject has radiotherapy or major surgery within 4 weeks prior to first dose of study drug.
* Subject has had chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 2 weeks prior to first dose of study drug.
* Subject has known hypersensitivity to EV or to any excipient contained in the drug formulation of EV; OR subject has known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells.
* Subject has known hypersensitivity to the following: docetaxel or to any of the other excipients listed in product label, including polysorbate 80, paclitaxel or to any of the other excipients listed in product label, such as macrogolglycerol ricinoleate 35 (Ph.Eur.); and vinflunine or to any of the other excipients listed in product label such as other vinca alkaloids (vinblastine,vincristine, vindesine, vinorelbine).
* Subject has known active keratitis or corneal ulcerations.
* Subject has other underlying medical condition that would impair the ability of the subject to receive or tolerate the planned treatment and follow-up.
* History of uncontrolled diabetes mellitus within 3 months of the first dose of study drug. Uncontrolled diabetes is defined as hemoglobin A1C (HbA1c) ≥ 8% or HbA1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.

Exclusion Criteria for COE

* Subject will be excluded from participation in the COE if they meet any of the exclusion criteria listed in the main protocol or if any of the following apply when the patient is evaluated for eligibility to participate in the COE portion of the study:
* Subject has been diagnosed with a new malignancy while on Arm B in the EV-301 study. Subjects with nonmelanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Subject has already started commercial EV or arrangements have been made for subject to start commercial EV which is reimbursed in their country. Additionally, if EV is commercially available with reimbursement in the potential subject's country, the subject can consider transitioning to the commercial product unless otherwise discussed with sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2025-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (158):
- United States (25):
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - University of California, Sacramento, California
  - Innovative Clinical Research, Whittier, California
  - University of Colorado, Denver, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, Lake Success, New York
  - Sidney Kimmel Center for Prostate and Urologic Cancers, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - White Plains Hospital Center for Cancer Care - Oncology Site, White Plains, New York
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Providence Portland Med Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Lifespan Rhode Island Hospital, Providence, Rhode Island
  - Saint Francis Hospital, Greenville, South Carolina
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Site AR54001, Buenos Aires, Argentina
- Australia (4):
  - Site AU61006, Adelaide
  - Site AU61001, Miranda
  - Site AU61004, St Leonards
  - Site AU61002, Sydney
- Austria (3):
  - Site AT43005, Linz
  - Site AT43001, Salzburg
  - Site AT43004, Vienna
- Belgium (9):
  - Site BE32011, Aalst
  - Site BE32007, Brussels
  - Site BE32013, Brussels
  - Site BE32010, Charleroi
  - Site BE32001, Ghent
  - Site BE32008, Ghent
  - Site BE32005, Hasselt
  - Site BE32003, Leuven
  - Site BE32009, Liège
- Canada (11):
  - Site CA15015, Calgary
  - Site CA15012, Edmonton
  - Site CA15014, London
  - Site CA15002, Montreal
  - Site CA15007, Montreal
  - Site CA15011, Oshawa
  - Site CA15004, Québec
  - Site CA15008, Saskatoon
  - Site CA15001, Sherbrooke
  - Site CA15005, Toronto
  - Site CA15013, Vancouver
- Denmark (3):
  - Site DK45003, Aalborg
  - Site DK45004, Copenhagen
  - Site DK45001, Herlev
- France (14):
  - Site FR33021, Besançon
  - Site FR33009, Bordeaux
  - Site FR33018, Bordeaux
  - Site FR33001, Brest
  - Site FR33016, Caen
  - Site FR33015, Lyon
  - Site FR33014, Marseille
  - Site FR33003, Nice
  - Site FR33022, Paris
  - Site FR33005, Pierre-Bénite
  - Site FR33004, Saint-Mandé
  - Site FR33002, Strasbourg
  - Site FR33019, Toulouse
  - Site FR33006, Villejuif
- Germany (5):
  - Site DE49011, Essen
  - Site DE49008, Heidelberg
  - Site DE49010, Münster
  - Site DE49003, Tübingen
  - Site DE49009, Würzburg
- Italy (7):
  - Site IT39008, Arezzo
  - Site IT39019, Cremona
  - Site IT39010, Milan
  - Site IT39025, Modena
  - Site IT39013, Pisa
  - Site IT39014, Reggio Emilia
  - Site IT39004, Terni
- Japan (25):
  - Site JP81010, Hirosaki, Aomori
  - Site JP81014, Kashiwa, Chiba
  - Site JP81007, Sapporo, Hokkaido
  - Site JP81026, Sapporo, Hokkaido
  - Site JP81020, Tsukuba, Ibaraki
  - Site JP81018, Morioka, Iwate
  - Site JP81009, Kita-gun, Kagawa-ken
  - Site JP81002, Yokohama, Kanagawa
  - Site JP81005, Sendai, Miyagi
  - Site JP81016, Sayama, Osaka
  - Site JP81024, Takatsuki, Osaka
  - Site JP81008, Bunkyo-ku, Tokyo
  - Site JP81012, Koto-ku, Tokyo
  - Site JP81013, Shinjuku-ku, Tokyo
  - Site JP81011, Ube, Yamaguchi
  - Site JP81015, Chiba
  - Site JP81019, Fukuoka
  - Site JP81023, Fukuoka
  - Site JP81004, Hiroshima
  - Site JP81001, Kyoto
  - Site JP81017, Niigata
  - Site JP81003, Okayama
  - Site JP81022, Osaka
  - Site JP81021, Tokushima
  - Site JP81006, Toyama
- Netherlands (4):
  - Site NL31002, Amsterdam
  - Site NL31003, Amsterdam
  - Site NL31009, Nijmegen
  - Site NL31001, Tilburg
- Portugal (3):
  - Site PT35102, Lisbon
  - Site PT35105, Lisbon
  - Site PT35106, Porto
- Russia (4):
  - Site RU70002, Ivanovo
  - Site RU70009, Obninsk
  - Site RU70005, Omsk
  - Site RU70015, Vologda
- South Korea (11):
  - Site KR82006, Daejeon
  - Site KR82007, Goyang-si
  - Site KR82012, Hwasun-gun
  - Site KR82002, Incheon
  - Site KR82001, Seongnam-si
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82008, Seoul
  - Site KR82009, Seoul
  - Site KR82010, Seoul
  - Site KR82005, Shin
- Spain (15):
  - Site ES34010, Badajoz
  - Site ES34002, Badalona
  - Site ES34001, Barcelona
  - Site ES34012, Barcelona
  - Site ES34023, Barcelona
  - Site ES34014, Córdoba
  - Site ES34003, Madrid
  - Site ES34013, Madrid
  - Site ES34015, Madrid
  - Site ES34017, Madrid
  - Site ES34011, Manresa
  - Site ES34019, Pamplona
  - Site ES34005, Seville
  - Site ES34007, Valencia
  - Site ES34008, Valencia
- Switzerland (2):
  - Site CH41002, Bern
  - Site CH41001, Chur
- Taiwan (6):
  - Site TW88602, Kaohsiung City
  - Site TW88605, Kaohsiung City
  - Site TW88606, Taichung
  - Site TW88601, Tainan
  - Site TW88604, Taipei
  - Site TW88607, Taoyuan District
- United Kingdom (6):
  - Site GB44005, London
  - Site GB44006, London
  - Site GB44004, Metropolitan Borough of Wirral
  - Site GB44002, Sheffield
  - Site GB44011, Southampton
  - Site GB44013, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Rosenberg JE, Mamtani R, Sonpavde GP, Loriot Y, Duran I, Lee JL, Matsubara N, Vulsteke C, Castellano D, Sridhar SS, Pappot H, Gurney H, Bedke J, van der Heijden MS, Galli L, Keam B, Masumori N, Meran J, O'Donnell PH, Park SH, Grande E, Sengelov L, Uemura H, Skaltsa K, Campbell M, Matsangou M, Wu C, Hepp Z, McKay C, Powles T, Petrylak DP. Health-related Quality of Life in Patients with Previously Treated Advanced Urothelial Carcinoma from EV-301: A Phase 3 Trial of Enfortumab Vedotin Versus Chemotherapy. Eur Urol. 2024 Jun;85(6):574-585. doi: 10.1016/j.eururo.2024.01.007. Epub 2024 Feb 28. PMID 38418343
- [Derived] Powles T, Rosenberg JE, Sonpavde GP, Loriot Y, Duran I, Lee JL, Matsubara N, Vulsteke C, Castellano D, Wu C, Campbell M, Matsangou M, Petrylak DP. Enfortumab Vedotin in Previously Treated Advanced Urothelial Carcinoma. N Engl J Med. 2021 Mar 25;384(12):1125-1135. doi: 10.1056/NEJMoa2035807. Epub 2021 Feb 12. PMID 33577729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with locally advanced or metastatic urothelial cancer (mUC) who had received a platinum-containing chemotherapy and had experienced disease progression or relapse during or following treatment with programmed cell death protein-1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitors.
Pre-assignment Details: Participants were stratified by Eastern Cooperative Oncology Group Performance Status (ECOG PS) (0 vs 1), regions of the world Western EU vs US vs Rest of World) and liver metastasis (Yes vs No).
Groups:
- Enfortumab Vedotin 1.25mg/kg: Participants received 1.25 milligrams per kilogram (mg/kg) of body weight enfortumab vedotin by intravenous (IV) infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
- Chemotherapy: Participants received either 75 milligram per square meter (mg/m^2) docetaxel by IV infusion over approximately 1 hour or 320 mg/m^2 vinflunine by IV infusion over approximately 20 minutes or 175 mg/m^2 paclitaxel by IV infusion over approximately 3 hours on day 1 of every 21-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
Period: Overall Study
Arm/Group | Enfortumab Vedotin 1.25mg/kg | Chemotherapy
Started | 301 | 307
Treated | 296 | 291
Completed | 56 (Participants still on treatment as of data cut-off date 15-Jul-2020) | 22 (Participants still on treatment as of data cut-off date 15-Jul-2020)
Not Completed | 245 | 285
Not completed — Adverse Event | 42 | 46
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Progressive Disease | 177 | 180
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 15 | 27
Not completed — Physician Decision | 7 | 22
Not completed — Miscellaneous | 1 | 6

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were randomized.
Groups:
- Enfortumab Vedotin 1.25 mg/kg: Participants received 1.25 mg/kg of body weight enfortumab vedotin by IV infusion over approximately 30 minutes on days 1, 8 and 15 of every 28day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
- Chemotherapy: Participants received either 75 mg/m^2 docetaxel by IV infusion over approximately 1 hour or 320 mg/m^2 vinflunine by IV infusion over approximately 20 minutes or 175 mg/m^2 paclitaxel by IV infusion over approximately 3 hours on day 1 of every 21-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy | Total
Number analyzed (Participants) | 301 | 307 | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.52 (9.11) | 66.81 (9.93) | 66.67 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 75 | 138
  Male | 238 | 232 | 470
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 24 | 53
  Not Hispanic or Latino | 230 | 238 | 468
  Unknown or Not Reported | 42 | 45 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 97 | 103 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 159 | 155 | 314
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 43 | 46 | 89
ECOG PS [Number; unit: participants] — ECOG PS was measured on 6 point scale 0-Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature
  2. Ambulatory & capable of all self-care but unable to carry out any work activities.Up & about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. Dead Participants were categorized based on ECOG PS 0 or 1
  participants
    ECOG PS=0 | 120 | 124 | 244
    ECOG PS=1 | 181 | 183 | 364
Liver Metastasis [Number; unit: participants] — Participants were categorized based on liver metastasis (yes or no).
  participants
    Liver Metastasis=No | 208 | 212 | 420
    Liver Metastasis=Yes | 93 | 95 | 188
Region [Number; unit: participants] — Participants were categorized based on region western europe, US and rest of the world.
  participants
    Western Europe | 126 | 129 | 255
    United States | 43 | 44 | 87
    Rest of the World | 132 | 134 | 266

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the documented date of death from any cause. OS was analyzed using Kaplan-Meier estimates. Participants who were still alive at the time of data cutoff date were to be censored at the last known alive date or at the data cutoff date, whichever was earlier.
Time Frame: From randomization until the analysis cut-off date of 15-Jul-2020 (median OS follow-up was 11.10 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enfortumab Vedotin 1.25 mg/kg: Participants received 1.25 mg/kg of body weight enfortumab vedotin by IV infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 301 | 307
months | 12.88 [10.58 to 15.21] | 8.97 [8.05 to 10.74]
Statistical Analysis 1: Comparison: Enfortumab Vedotin 1.25 mg/kg vs Chemotherapy; Test type: Superiority; p = 0.00142, Stratified Log rank — Stratification factors were ECOG PS, geographic region and liver metastasis. P-value was based on log-rank test. P-value of overall survival is ≤ the predetermined 1-sided significance level of 0.00679 based on the number of observed deaths; Stratified Hazard Ratio = 0.702, 95% CI 2-sided [0.556 to 0.886] — Cox proportional hazards model with treatment, ECOG PS, geographic region and liver metastasis as the explanatory variables

2. Secondary Outcome: Progression Free Survival on Study Therapy (PFS1) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS: time from date of randomization until date of documented radiological disease progression (PD) per investigator based on RECIST V1.1, or until death due to any cause, whichever occurred first. PD: >= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression. A participant who neither progressed nor died was censored at date of last radiological assessment (RA)/ date of randomization if no post-baseline RA was available. Participants who received any further anticancer therapy (ACT) for disease before radiological progression was censored at date of last RA before ACT started and participants who had PD/death after >=2 missed RAs were censored at last RA prior to 2 or more missed RAs. Kaplan-Meier estimates was used. Median time of follow-up for PFS was based on data cut-off & is same as median follow-up time for OS.
Time Frame: From randomization until the analysis cut-off date of 15-Jul-2020 (median OS follow-up was 11.10 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 301 | 307
months | 5.55 [5.32 to 5.82] | 3.71 [3.52 to 3.94]
Statistical Analysis 1: Comparison: Enfortumab Vedotin 1.25 mg/kg vs Chemotherapy; Test type: Superiority; p < 0.00001, Stratified Log Rank — Stratification factors were ECOG PS, geographic region and liver metastasis. P-value was based on log-rank test. P value of PFS is ≤ the predetermined 1-sided significance level of 0.02189 based on the number of observed PFS events; Stratified Hazard Ratio = 0.615, 95% CI 2-sided [0.505 to 0.748] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR) as Per RECIST V1.1
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) based on the RECIST v1.1. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. ORR was analysed using exact method based on binomial distribution (Clopper-Pearson). Median time of follow up for ORR was based on data cut-off and is same as median follow-up time for OS.
Time Frame: From randomization until the analysis cut-off date of 15-Jul-2020 (median OS follow-up was 11.10 months)
Population: Response Evaluable Set (RES): The RES was defined as all participants in the FAS who had measurable disease (per RECIST v1.1) per investigator at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 288 | 296
percentage of participants | 40.6 [34.90 to 46.54] | 17.9 [13.71 to 22.76]
Statistical Analysis 1: Comparison: Enfortumab Vedotin 1.25 mg/kg vs Chemotherapy; Test type: Superiority; p < 0.001, Stratified Cochran-Mantel-Haenszel — "Stratification factors were ECOG PS, Region and Liver Metastasis

4. Secondary Outcome: Disease Control Rate (DCR) as Per RECIST V1.1
Description: DCR was defined as the percentage of participants with a CR, PR or a stable disease (SD) based on RECIST v1.1. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters while on study drug. Progressive disease is defined in PFS1 endpoint. DCR was analysed using exact method based on binomial distribution (Clopper-Pearson). Median time of follow up for DCR was based on data cut-off and is same as median follow-up time for OS.
Time Frame: From randomization until the analysis cut-off date of 15-Jul-2020 (median OS follow-up was 11.10 months)
Population: RES Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 288 | 296
percentage of participants | 71.9 [66.30 to 76.99] | 53.4 [47.52 to 59.17]
Statistical Analysis 1: Comparison: Enfortumab Vedotin 1.25 mg/kg vs Chemotherapy; Test type: Superiority; p < 0.001, Stratified Cochran-Mantel-Haenszel — Stratification factors were ECOG PS, Region and Liver Metastasis

5. Secondary Outcome: Duration of Response (DOR) as Per RECIST V1.1
Description: DOR: time from the date of the first CR/PR (whichever is first recorded) that was subsequently confirmed as assessed by investigator to the date of documented PD or death due to any cause whichever occurred first. If a participant has neither progressed nor died, the participant was censored at the date of last RA or at the date of first CR/PR if no subsequent post-baseline RA was available. Participants who received any further ACT for the disease before radiological progression were censored at the date of the last RA before the ACT started. In addition, participants who had PD/death after >= 2 missed RAs were censored at the last RA prior to the 2 or more missed RAs. Kaplan-Meier estimates was used. Median time of follow up for DOR was based on data cut-off and is same as median follow-up time for OS. CR/PR and PD were defined in ORR and PFS1 endpoints, respectively.
Time Frame: From date of first objective response until the analysis cut-off date of 15-Jul-2020 (median OS follow-up was 11.10 months)
Population: RES population with available data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 117 | 53
months | 7.39 [5.59 to 9.46] | 8.11 [5.65 to 9.56]

6. Secondary Outcome: Change From Baseline to Week 12 in European Organisation for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire Global Health Status (QL2 Score)
Description: EORTC QLQ-C30 is a generic questionnaire consisting of 30 items. The instrument yields functional scales (physical, role, emotional, cognitive, social), symptom scales/items (fatigue, Nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea), global health status, and financial impact score. Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). The recall period for each question is "during the past week". All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state. Higher scores on the global health status and functioning scales indicate better health status/function.
Time Frame: Baseline and week 12
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 127 | 102
score on a scale | -2.30 (18.02) | -5.72 (16.04)

7. Secondary Outcome: Change From Baseline to Week 12 in EuroQOL 5-dimension 5-level Questionnaire [EQ-5D-5L] Visual Analog Scale (VAS)
Description: EQ-5D-5L is a health status instrument for self-reported assessment of 5 domains of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is rated by selecting 1 of 5 standardized categorizations ranging from no problem to extreme problem. The final question is a visual analogue scale (VAS) to rank health status from 0 (best health imaginable) to 100 (worst health imaginable).
Time Frame: Baseline and week 12
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 124 | 102
score on a scale | -1.8 (16.6) | -5.3 (14.5)

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A TEAE is defined as an AE observed or worsened after starting administration of the study drug.
Time Frame: From first dose up to 30 days after last dose (Median (range) time on study drug was 4.99 (0.5, 19.4) months in enfortumab vedotin and 3.45 (0.2, 15.0) months in chemotherapy group)
Population: The safety analysis set (SAF) consisted of all participants who received any amount of study drug, and was used for safety analyses.
Measure: Number; unit: participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 296 | 291
participants | 290 | 288

9. Secondary Outcome: Number of Participants With ECOG Performance Status
Description: ECOG performance status was measured on an 6 point scale. 0-Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead. Number of participants with ECOG PS was reported.
Time Frame: End of treatment (EOT) (Median (range) time on study drug was 4.99 (0.5, 19.4) months in enfortumab vedotin and 3.45 (0.2, 15.0) months in chemotherapy group)
Population: Safety population with available data.
Measure: Number; unit: participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg | Chemotherapy
Number analyzed (Participants) | 184 | 219
participants
  ECOG PS = 0 | 34 | 57
  ECOG PS = 1 | 110 | 118
  ECOG PS >1 | 40 | 44

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose (Median (range) time on study drug was 4.99 (0.5, 19.4) months in enfortumab vedotin and 3.45 (0.2, 15.0) months in chemotherapy group)
Groups:
- Enfortumab Vedotin: Participants received 1.25 mg/kg of body weight enfortumab vedotin by IV infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
Arm/Group | Enfortumab Vedotin | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 130/296 | 161/291
Serious Adverse Events (participants affected / at risk) | 138/296 | 128/291
Other Adverse Events (participants affected / at risk) | 284/296 | 266/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin (N=296) | Chemotherapy (N=291)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (7)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 16 (16)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 8 (9)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 4 (6)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 2 (2)
General physical health deterioration (General disorders) | 2 (3) | 5 (5)
Malaise (General disorders) | 2 (2) | 3 (4)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 9 (11)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (4) | 1 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Abscess bacterial (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 2 (4)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (2) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (2)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (5)
Pneumonia (Infections and infestations) | 12 (14) | 7 (9)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (3)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (5)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (6) | 3 (5)
Septic shock (Infections and infestations) | 4 (6) | 1 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (7) | 6 (7)
Urinary tract infection bacterial (Infections and infestations) | 9 (10) | 3 (3)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 6 (7)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 5 (6)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (15) | 7 (7)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Frontotemporal dementia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 19 (31) | 7 (7)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Choluria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 5 (6) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Vascular compression (Vascular disorders) | 0 (0) | 1 (1)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin (N=296) | Chemotherapy (N=291)
Anaemia (Blood and lymphatic system disorders) | 57 (98) | 83 (136)
Neutropenia (Blood and lymphatic system disorders) | 16 (30) | 20 (37)
Dry eye (Eye disorders) | 19 (24) | 3 (3)
Lacrimation increased (Eye disorders) | 30 (37) | 12 (15)
Vision blurred (Eye disorders) | 16 (20) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 37 (52) | 24 (33)
Constipation (Gastrointestinal disorders) | 81 (116) | 72 (105)
Diarrhoea (Gastrointestinal disorders) | 98 (171) | 64 (89)
Dry mouth (Gastrointestinal disorders) | 24 (26) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 19 (22) | 9 (10)
Nausea (Gastrointestinal disorders) | 89 (119) | 73 (92)
Stomatitis (Gastrointestinal disorders) | 27 (35) | 19 (27)
Vomiting (Gastrointestinal disorders) | 38 (50) | 44 (57)
Asthenia (General disorders) | 43 (85) | 39 (85)
Chills (General disorders) | 16 (18) | 5 (5)
Fatigue (General disorders) | 107 (197) | 77 (121)
Malaise (General disorders) | 12 (13) | 19 (24)
Oedema peripheral (General disorders) | 25 (32) | 39 (46)
Pyrexia (General disorders) | 60 (99) | 33 (47)
Conjunctivitis (Infections and infestations) | 18 (23) | 2 (2)
Nasopharyngitis (Infections and infestations) | 15 (18) | 9 (9)
Urinary tract infection (Infections and infestations) | 21 (22) | 12 (15)
Fall (Injury, poisoning and procedural complications) | 15 (19) | 8 (8)
Alanine aminotransferase increased (Investigations) | 27 (45) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 36 (56) | 5 (7)
Blood creatinine increased (Investigations) | 26 (38) | 6 (6)
Lymphocyte count decreased (Investigations) | 12 (35) | 17 (50)
Neutrophil count decreased (Investigations) | 32 (70) | 52 (159)
Weight decreased (Investigations) | 47 (73) | 20 (20)
White blood cell count decreased (Investigations) | 16 (45) | 32 (97)
Decreased appetite (Metabolism and nutrition disorders) | 119 (157) | 78 (104)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (64) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (22) | 10 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 (28) | 8 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (36) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (23) | 36 (44)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (28) | 23 (25)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (23) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (23) | 31 (40)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (20) | 13 (19)
Dizziness (Nervous system disorders) | 26 (34) | 16 (18)
Dysgeusia (Nervous system disorders) | 74 (99) | 23 (28)
Headache (Nervous system disorders) | 9 (10) | 17 (22)
Neuropathy peripheral (Nervous system disorders) | 20 (45) | 16 (20)
Paraesthesia (Nervous system disorders) | 15 (23) | 8 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 102 (301) | 66 (99)
Insomnia (Psychiatric disorders) | 31 (32) | 23 (25)
Haematuria (Renal and urinary disorders) | 31 (41) | 22 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 17 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 26 (36)
Alopecia (Skin and subcutaneous tissue disorders) | 139 (163) | 110 (121)
Drug eruption (Skin and subcutaneous tissue disorders) | 26 (40) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 50 (57) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 102 (153) | 20 (20)
Rash (Skin and subcutaneous tissue disorders) | 49 (77) | 16 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 49 (99) | 6 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 19 (20) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03474107/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03474107/SAP_001.pdf